CLINICAL TRIAL: NCT02616653
Title: Identification of the L3-L4 Intervertebral Space in Obese Parturients at Term in the Sitting and Lateral Positions: Manual Palpation (Tuffier's Line Method) Versus Ultrasound Imaging
Brief Title: Identification of the L3-L4 Intervertebral Space in Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 15.251
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Pregnancy; Obesity; Obstetrical Anesthesia
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitting followed by lateral position (Active Comparator): First half of participants will be assigned to have their L3-L4 intervertebral space located first in the sitting position followed by the lateral position using the palpation method confirmed by US. (L3-L4 location: Palpation method confirmed by US)
  Interventions: Procedure: L3-L4 location: Palpation method confirmed by US
- Lateral followed by sitting position (Active Comparator): Second half of participants will be assigned to have their L3-L4 intervertebral space located first in the lateral position followed by the sitting position using the palpation method confirmed by US. (L3-L4 location: Palpation method confirmed by US)
  Interventions: Procedure: L3-L4 location: Palpation method confirmed by US

INTERVENTIONS:
Procedure: L3-L4 location: Palpation method confirmed by US — An anesthesiologist will locate the L3-L4 space using the palpation method (Tuffier's line). An investigator trained in US imaging will proceed to the US exam of the spine specifically aiming to identify the L3-L4 intervertebral space. The investigator will note if the same level was identified and if not, which one was according to the US exam.

SUMMARY:
This study is designed to determine the frequency of Tuffier's line overestimation (2 lumbar levels or more) when the palpation method is used in obese parturients at term in the lateral position compared to the sitting position.

Hypothesis: The L3-L4 intervertebral space identified by the palpation method will be two levels higher than the level determined by ultrasonography (US) more often in the lateral than in the sitting position.

DETAILED DESCRIPTION:
For years now, anesthesiologists have used anatomical landmarks to guide neuraxial anesthesia and analgesia techniques in obstetric patients. Traditionally, Tuffier's line (intercristal line) has been used as a reference and corresponds to a horizontal line drawn between the upper part of the iliac crests that is thought to intersect the spine at the level of the L4 spinous process or the L4-L5 intervertebral space. However, many studies have found this anatomical landmark to be unreliable reporting the Tuffier's line to intersect the spine at levels ranging from the L3-L4 to L5-S1 intervertebral spaces. Regarding the obstetrical population, the anatomical position of the Tuffier's line was found to be even higher presumably due to the exaggerated lordosis of pregnancy.

Neuraxial techniques used for obstetrical anesthesia and analgesia include epidurals, spinals and combined epidural-spinal (CSE) techniques. The correct identification of the intervertebral space for neuraxial analgesia and anesthesia is very important especially if using a spinal injection such as is done when performing a CSE.

Neuraxial techniques can be done in the sitting or the lying lateral position. When expecting a more challenging technique, such as in an obese patient, anesthesiologists will usually choose to perform the technique with patients in the sitting position. But the lateral position is preferred in certain conditions such as in premature rupture of membranes where there is a risk of umbilical cord prolapse, in women experiencing a vasovagal response caused by the needle insertion or upon assuming the sitting position, or because of the anesthesiologist's preference.

US-guided regional techniques are gaining popularity both for the general population as well as for the pregnant women. It has been shown to be a more reliable tool than the palpation method in identifying a specific lumbar intervertebral level. The use of US imaging for neuraxial techniques in pregnant women has been shown to reduce the numbers of attempts, improve the comfort of the patient during the procedure and increase the precision in identifying the intervertebral space at which the technique is being performed. Obesity can make regional techniques extremely challenging and US imaging becomes a valuable tool in this setting.

Methods:

Participants will be positioned on an exam table in the sitting position for the first half of the group and the lateral position for the other half. For the sitting position, the participants will have both feet supported by a foot rest while being asked to round back by lowering their head on their chest and pushing out their back to assume a fetal like position. If necessary, the women may be asked to hold a pillow to improve their position to get the ideal conditions for the palpation of the Tuffier's line and intervertebral spaces. For the lateral position, the participants will be placed on the left lateral side with flexion of the knees and hip, and flexion of the head and neck with a pillow supporting them. Again, the women will be instructed to adopt a fetal position by rounding their back.

An anesthesiologist who is assigned to the obstetrical floor for the day and who is not an investigator in this study will be asked to perform the palpation method. He/she will proceed with the identification of the Tuffier's line (upper part of the iliac crests) and determine the level of intersection with the spine. This anatomical landmark will then be used to estimate the location of the L3-L4 intervertebral space which is the space frequently chosen to proceed to a neuraxial technique. Once the level is identified, it will be marked and hidden under a hypoallergenic paper tape. The anesthesiologist will then leave the room while the investigator trained in US imaging will proceed to the US exam of the spine specifically aiming to identify the L3-L4 intervertebral space. Once located, the investigator will be able to look at the skin mark made by the anesthesiologist and compare it to the level he/she will have determined to be at the L3-L4 level by US imaging. The investigator will note if the same level was identified and if not, which one was according to the US exam. The paper tape will be reapplied over the lumbar spine to mask any anatomical marks (birth marks or scars) that may influence the anesthesiologist who will be asked to step in again to proceed to the palpation method in the other position, again marking the area which he/she thinks corresponds to the L3-L4 space. US imaging will be repeated in the second position and the level obtained by the exam will be compared to the one obtained by the palpation method in the same way as the first position. The investigators expect the total time for the procedure to be of 20-30 minutes. Participants will be asked to rate their level of comfort during the procedure in both positions using a verbal rating scale from 0 to 10.

ELIGIBILITY:
Inclusion Criteria:

* Obese pregnant women (BMI equal or superior to 30)
* Pregnancy at term (37 weeks or more)

Exclusion Criteria:

* American Society of Anesthesiologists' physical status of 4 or 5
* Scoliosis or any other anomaly of the spine
* Prior spine surgery
* Inability to assume the correct position due to back pain
* Inability to collaborate
* Labouring women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Estimation of Tuffier's line using the palpation method | On Day one during medical appointment at the obstetrics clinic
  Incidence of overestimation of the Tuffier's line (2 lumbar levels or more) using the palpation method in the sitting position compared to the lateral position

SECONDARY OUTCOMES:
Impact of fundal height on estimation of the Tuffier's line using the palpation method | On Day one during medical appointment at the obstetrics clinic
  Impact of fundal height on overestimation of the Tuffier's line using the palpation method in the sitting position compared to the lateral position
Comfort level using a verbal rating scale | On Day one during medical appointment at the obstetrics clinic
  Level of comfort during the procedure in the sitting and lateral positions using a verbal rating scale (0 being totally comfortable, 10 totally uncomfortable)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Garneau, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No